CLINICAL TRIAL: NCT00365417
Title: A Phase II Clinical Trial of Bevacizumab Beginning Concurrently With a Sequential Regimen of Doxorubicin and Cyclophosphamide Followed by Docetaxel and Capecitabine as Neoadjuvant Therapy Followed by Postoperative Bevacizumab Alone for Women With Locally Advanced Breast Cancer
Brief Title: Therapy With Bevacizumab (BEV), Doxorubicin, and Cyclophosphamide Followed by BEV, Docetaxel, and Capecitabine Before Surgery Followed by BEV Alone After Surgery for Women With Locally Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Collaborators: Genentech, Inc. (Industry); Hoffmann-La Roche (Industry); International Drug Development Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSABP FB-4
Record Dates: First submitted 2006-08-15; First posted 2006-08-17 (Estimated); Results first posted 2010-08-12 (Estimated); Last update posted 2021-04-13 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer
Keywords: NSABP; Doxorubicin; Cyclophosphamide; Bevacizumab; Capecitabine; Docetaxel; Breast cancer; Locally advanced; Neoadjuvant; Locally advanced breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Doxorubicin; Cyclophosphamide; Capecitabine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Doxorubicin+Cyclophosphamide+Bevacizumab (Experimental)
  Interventions: Drug: Bevacizumab; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Capecitabine; Drug: Docetaxel

INTERVENTIONS:
Drug: Bevacizumab — 15 mg/kg IV every 21 days x 4 cycles, then after clinical response assessment, 15 mg/kg IV every 21 days x 2 cycles, then following surgery, 15 mg/kg every 21 days x 10 cycles
  Other Names: Avastin
Drug: Doxorubicin — 60 mg/m^2 IV every 21 days x 4 cycles
Drug: Cyclophosphamide — 600 mg/m^2 IV every 21 days x 4 cycles
Drug: Capecitabine — Following clinical response assessment, 650 mg/m^2 twice a day (orally), days 1-14 every 21 days x 4 cycles
  Other Names: Xeloda
Drug: Docetaxel — Following clinical response assessment, 75 mg/m^2 IV every 21 days x 4 cycles
  Other Names: Taxotere

SUMMARY:
Bevacizumab is an angiogenesis inhibitor which means it works to stop blood vessel formation in tumors. Without new blood vessels, the growth of a tumor is slowed. Chemotherapy drugs kill cancer cells more directly. This study will evaluate:

* How bevacizumab, given with chemotherapy before surgery, and then bevacizumab given alone after surgery, will affect locally advanced breast tumors
* Side effects from adding bevacizumab to chemotherapy
* Whether adding bevacizumab to chemotherapy for breast cancer will affect the heart
* If receiving bevacizumab will have any effect on how patients recover from surgery
* Side effects of the combinations of drugs used in this study

DETAILED DESCRIPTION:
Initial trials of neoadjuvant chemotherapy administered for locally advanced tumors, including those in breast cancer, demonstrated therapy could induce sufficient tumor regression to allow for the resection of otherwise unresectable tumors. Subsequent demonstration of the equivalence of lumpectomy to mastectomy in patients with operable breast cancer, stimulated interest in the concept of using preoperative chemotherapy to reduce large, but operable, primary tumors to allow for lumpectomy in women who would otherwise require a mastectomy. Given the data from previous studies, it is appropriate to continue development of sequential doxorubicin/cyclophosphamide/docetaxel regimens to improve on clinical and pathologic response rates. FB-4 is a Phase II, single arm study for women with locally advanced human epidermal growth factor receptor 2 (HER2)-negative breast cancer diagnosed by core needle biopsy. The primary aim of the study is to determine the pathologic complete response rate in the breast following neoadjuvant chemotherapy combined with bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be female.
* The patient must be greater than/equal to 18 years old
* The diagnosis of invasive adenocarcinoma of the breast must have been made by core needle biopsy or limited incisional biopsy.
* Patients must have clinical Stage IIIA, IIIB, or IIIC disease (American Joint Committee on Cancer [AJCC] staging criteria) with a primary breast tumor that is greater than/equal to 2.0 cm measured by clinical exam, unless the patient has inflammatory breast carcinoma, in which case measurable disease is not required.
* Patients must have the ability to swallow oral medication.
* The patient's Eastern Cooperative Oncology Group (ECOG) performance status must be 0 or 1.
* At the time of study entry, blood counts must meet the following criteria:

  * Absolute neutrophil count (ANC) must be greater than/equal to 1200/mm3.
  * Platelet count must be greater than/equal to 100,000/mm^3.
  * Hemoglobin must be greater than/equal to 10 g/dL.
* The following criteria for evidence of adequate hepatic function must be met:

  * total bilirubin must be less than/equal to upper limit of normal (ULN) for the lab unless the patient has a grade 1 bilirubin elevation (greater than ULN to 1.5 x ULN) due to Gilbert's disease or similar syndrome involving slow conjugation of bilirubin; and
  * alkaline phosphatase must be less than 2.5 x ULN for the lab; and
  * aspartate aminotransferase (AST) must be less than/equal to 1.5 x ULN for the lab.
  * Alkaline phosphatase and AST may not both be greater than the ULN. For example, if the alkaline phosphatase is greater than the ULN but less than/equal to 2.5 x ULN, then the AST must be less than/equal to the ULN. If the AST is greater than the ULN but less than/equal to 1.5 x ULN, then the alkaline phosphatase must be less than/equal to ULN.
* Patients with either skeletal pain or alkaline phosphatase that is greater than ULN but less than/equal to 2.5 x ULN are eligible for inclusion in the study if a bone scan or positron emission tomography (PET) scan does not demonstrate metastatic disease. Patients with suspicious findings on bone scan or PET scan are eligible if suspicious findings are confirmed as benign by x-ray, magnetic resonance imaging (MRI), or biopsy.
* Patients with AST or alkaline phosphatase greater than ULN are eligible for inclusion in the study if liver imaging (computed tomography [CT], MRI, or PET scan) does not demonstrate metastatic disease and adequate hepatic function.
* The following criteria for evidence of adequate renal function must be met:

  * Serum creatinine less than/equal to ULN for the lab.
  * Calculated creatinine clearance must be greater than 50 mL/min.
* Urine protein/creatinine (UPC) ratio must be less than 1.0.
* Patients must have their left ventricular ejection fraction (LVEF) assessed by multigated acquisition (MUGA) scan or echocardiogram within 3 months prior to study entry. The LVEF must be greater than/equal to the lower limit of normal (LLN) for the cardiac imaging facility performing the MUGA scan or echocardiogram. Note: If the cardiac imaging facility cannot provide a LLN, use 50% as the LLN value.

Note: Since the pre-entry LVEF serves as the baseline for comparing subsequent LVEF assessments to determine if bevacizumab therapy can be continued following doxorubicin and cyclophosphamide (AC) and postoperatively, it is critical that this baseline study be an accurate assessment of the patient's LVEF. If the baseline LVEF is greater than 65%, the MUGA scan or echocardiogram must be repeated prior to study entry. The lower of the two LVEF values should be used as the baseline LVEF.

* Patients must have an electrocardiogram (EKG) within 3 months prior to study entry.

Exclusion Criteria:

* Tumor determined to be strongly HER2-positive by immunohistochemistry (3+) or by fluorescent in situ hybridization (positive for gene amplification).
* Excisional biopsy for this primary tumor.
* Synchronous bilateral invasive breast cancer.
* Surgical axillary staging procedure prior to study entry (Exceptions: 1) fine needle aspiration (FNA) of an axillary node is permitted for any patient, and 2) although not recommended, a sentinel lymph node biopsy for patients with clinically negative axillary nodes is permitted.)
* History of any of the following cancers:

  * Ipsilateral breast cancer: invasive, ductal carcinoma in situ (DCIS) treated with any therapy other than excision
  * Contralateral breast cancer: invasive within the past 5 years (Patients with history of DCIS or synchronous DCIS are eligible)
  * History of non-breast malignancies within the 5 years prior to study entry. Patients with the following cancers are eligible if diagnosed and treated within the previous 5 years: carcinoma in situ of the cervix, carcinoma in situ of the colon, melanoma in situ, and basal cell and squamous cell carcinoma of the skin.
* Prior therapy with anthracyclines, taxanes, capecitabine, or bevacizumab for any malignancy.
* Treatment including radiation therapy, chemotherapy, biotherapy, and/or hormonal therapy administered for the currently diagnosed breast cancer prior to study entry. The only exception is hormonal therapy, which may have been given for up to a total of 28 days anytime after diagnosis and before study entry. In such a case, hormonal therapy must stop at or before study entry and be re-started, if indicated, following chemotherapy.
* Any of the following cardiac conditions:

  * angina pectoris that requires the use of anti-anginal medication;
  * history of documented congestive heart failure;
  * serious cardiac arrhythmia requiring medication;
  * severe conduction abnormality;
  * valvular disease with documented cardiac function compromise; or
  * uncontrolled hypertension defined as blood pressure greater than 150/90 on antihypertensive therapy. (Patients with hypertension that is well controlled on medication are eligible.)
* History of myocardial infarction documented by elevated cardiac enzymes or persistent regional wall abnormalities on assessment of left ventricular (LV) function.
* History of transient ischemic attack (TIA) or cerebrovascular accident (CVA).
* History of other arterial thrombotic event within 12 months before study entry.
* Symptomatic peripheral vascular disease.
* Any significant bleeding within 6 months before study entry.
* Serious or non-healing wound, skin ulcers, or bone fracture.
* Gastroduodenal ulcer(s) determined by endoscopy to be active.
* Invasive procedures defined as follows:

  * Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to planned start of study therapy. (Note: Placement of a vascular access device is not considered a major surgical procedure.)
  * Anticipation of need for major surgical procedures (other than the required breast surgery) during the course of the study.
* Known bleeding diathesis or coagulopathy. (Patients on warfarin with an in-range international normalized ratio [INR] [usually between 2 and 3] are eligible.)
* Other nonmalignant systemic disease (cardiovascular, renal, hepatic, diabetes, etc.) that would preclude the patient from receiving study treatment or would prevent required follow-up.
* Sensory/motor neuropathy greater than/equal to grade 2, as defined by the NCI's Common Terminology Criteria for Adverse Events Version 3.0 (CTCAE v3.0).
* Conditions that would prohibit administration of corticosteroids.
* History of hypersensitivity reaction to drugs formulated with polysorbate 80.
* Therapy with any hormonal agent such as raloxifene, tamoxifen, or other selective estrogen receptor modulator (SERM), either for osteoporosis or breast cancer prevention. Patients are eligible only if these medications are discontinued prior to study entry.
* Any sex hormonal therapy, e.g., birth control pills, ovarian hormonal replacement therapy, etc. These patients are eligible if this therapy is discontinued prior to study entry. (Women of reproductive potential must agree to use an effective non-hormonal method of contraception during study therapy and for at least 3 months after completion of bevacizumab.)
* Pregnancy or lactation at the time of study entry.
* Use of any investigational agent within 4 weeks prior to enrollment in the study.
* Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-08; Primary Completion 2008-02 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (1):
- NSABP Foundation, Inc., Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemo Plus Bevacizumab: Bevacizumab beginning concurrently with a sequential regimen of doxorubicin and cyclophosphamide followed by docetaxel and capecitabine as neoadjuvant therapy followed by postoperative bevacizumab alone for women with HER2 negative locally advanced breast cancer
Period: Overall Study
Arm/Group | Chemo Plus Bevacizumab
Started | 45
Completed | 45
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Chemo Plus Bevacizumab
Number analyzed (Participants) | 45
Age, Customized [Number; unit: participants]
  18 to less than 50 years | 19
  Between 50 and 59 years | 13
  Greater than 59 years | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 43
  Black or African American | 1
  Native Hawaiian or other Pacific Islander | 0
  American Indian or Alaskan Native | 0
  Asian | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 42

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response (pCR) in the Breast
Description: Measured by no histologic evidence of invasive tumor cells in the surgical breast specimen
Time Frame: Approximately 7 months
Measure: Number; unit: participants
Groups:
- Neoadjuvant Study Treatment: Doxorubicin, cyclophosphamide, and bevacizumab followed by docetaxel and capecitabine
Arm/Group | Neoadjuvant Study Treatment
Number analyzed (Participants) | 45
participants
  pCR in the breast | 4
  No pCR in the breast | 38
  No data available | 3

2. Secondary Outcome: pCR in the Breast and Nodes
Description: Measured by no histologic evidence of invasive tumor cells in the surgical breast specimen, axillary nodes, or sentinel nodes
Time Frame: Approximately 7 months
Measure: Number; unit: participants
Arm/Group | Neoadjuvant Study Treatment
Number analyzed (Participants) | 45
participants
  pCR in the breast and nodes | 4
  No pCR in the breast and nodes | 38
  No data available | 3

3. Secondary Outcome: Clinical Response Rate (cRR) of the Sequential Regimen
Description: Clinical tumor measurements were required before study entry & before cycle 5 of chemotherapy (between AC & TX). Final tumor measurements were obtained 4-5 weeks after the last dose of chemotherapy. Clinical tumor assessments by physical examination were recommended before each chemotherapy cycle. The criteria proposed by the Response Evaluation Criteria in Solid Tumors Committee(RECIST) were used to define clinical response status. CR was defined as the disappearance of all lesions with no evidence of PD. PR was defined as at least 30% decrease in the sum of the longest diameter of target lesions, using as reference the baseline sum longest diameter and/or the persistence of greater than or equal to 1 nontarget lesion without worsening of any other clinical manifestations of disease. PD was defined as at least a 20% increase in the sum of the longest diameter of target lesions, the appearance of new lesions, or unequivocal progression of existing lesions.
Time Frame: Approximately 6 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Chemo Plus Bevacizumab
Number analyzed (Participants) | 45
percentage of patients | 77.27 [62.16 to 88.53]

4. Secondary Outcome: Reported Adverse Events
Description: Number of Adverse Events
Time Frame: Approximately 14 months
Measure: Number; unit: events
Arm/Group | Neoadjuvant Study Treatment
Number analyzed (Participants) | 45
events | 566

5. Secondary Outcome: Cardiac Events
Description: Events: Congestive Heart Failure; Cardiac Death
Time Frame: Assessments throughout; up to 18 months following study entry
Population: Symptomatic cardiac toxicity was not observed in this study.
Measure: Number; unit: cardiac events
Arm/Group | Chemo Plus Bevacizumab
Number analyzed (Participants) | 45
cardiac events | 0

6. Secondary Outcome: Progression-free Survival
Description: Percentage of patients free from disease progression. Progression is determined using international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee. At least a 20% increase in the sum of the longest diameter of the target lesions. Other manifestations of progressive disease would also be classified as disease progression, eg., appearance of one or more new lesions in the breast, regional lymph nodes or distant sites, unequivocal progression of existing non-target lesions, and appearance of inflammatory carcinoma on clinical exam.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Chemo Plus Bevacizumab
Number analyzed (Participants) | 45
percentage of patients | 57.69 [42 to 70.56]

7. Secondary Outcome: Overall Survival
Description: Percentage of patients alive.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Chemo Plus Bevacizumab
Number analyzed (Participants) | 45
percentage of patients | 74.52 [58.5 to 85.09]

8. Secondary Outcome: Number of Patients With at Least One Surgical Complications (Wound Dehiscence, Infection, Seroma, or Hematoma).
Description: Number of patients with at least one surgical complications (wound dehiscence, infection, seroma, or hematoma)
Time Frame: Two (2) years
Population: Of the 45 patients, 43 patients had surgery and therefore 43 patients in this outcome.
Measure: Number; unit: participants
Arm/Group | Chemo Plus Bevacizumab
Number analyzed (Participants) | 43
participants | 24

ADVERSE EVENTS:
Time Frame: Assessments throughout up to 3 years, 3 months
Arm/Group | Chemo Plus Bevacizumab
Serious Adverse Events (participants affected / at risk) | 14/45
Other Adverse Events (participants affected / at risk) | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemo Plus Bevacizumab (N=45)
Diarrhea (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
Hand-foot (Skin and subcutaneous tissue disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Infection - blood (Infections and infestations) | 1
Infection - catheter related (Infections and infestations) | 1
Infection - lung (pneumonia) (Infections and infestations) | 2
Infection - skin (cellulites) (Infections and infestations) | 3
Infection - ungual (nails) (Infections and infestations) | 1
Infection - urinary tract NOS (Infections and infestations) | 1
Infection with normal ANC - sinus (Infections and infestations) | 1
Infection with normal ANC - skin (cellulites) (Infections and infestations) | 2
Infection with normal ANC - upper airway NOS (Infections and infestations) | 1
Infection with normal ANC - urinary tract NOS (Infections and infestations) | 1
Infection with normal ANC - wound (Infections and infestations) | 1
Insomnia (General disorders) | 1
Mucositis (clinical exam) - oral cavity (Gastrointestinal disorders) | 1
Mucositis (functional/symptomatic) - esophagus (Gastrointestinal disorders) | 1
Mucositis (functional/symptomatic) - oral cavity (Gastrointestinal disorders) | 2
Pain - abdominal NOS (General disorders) | 2
Pain - back (General disorders) | 1
Pain - musculoskeletal (hip) (General disorders) | 1
Syncope (fainting) (General disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chemo Plus Bevacizumab (N=45)
ALT (Investigations) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 35
Anorexia (General disorders) | 15
Blood - other HCT (Investigations) | 5
Constipation (Gastrointestinal disorders) | 6
Cytokine release syndrome (General disorders) | 4
Dehydration (Gastrointestinal disorders) | 9
Dermatitis - radiation (Skin and subcutaneous tissue disorders) | 9
Diarrhea (Gastrointestinal disorders) | 15
Dizziness (Nervous system disorders) | 3
Dysphagia (Gastrointestinal disorders) | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Fatigue (General disorders) | 32
Febrile neutropenia (Infections and infestations) | 11
Hand-foot (Skin and subcutaneous tissue disorders) | 26
Heartburn (Gastrointestinal disorders) | 9
Hemaglobin (Blood and lymphatic system disorders) | 12
Hemorrhoids (Gastrointestinal disorders) | 4
Hot flashes (Endocrine disorders) | 11
Hyperglycemia (Investigations) | 4
Hypertension (Cardiac disorders) | 11
Hypocalcemia (Investigations) | 3
Hypokalemia (Investigations) | 4
Hypophosphatemia (Investigations) | 3
Infection (documented clincally) - upper airway NOS (Infections and infestations) | 3
Infection - bladder (urinary) (Infections and infestations) | 4
Infection - other (thrush) (Infections and infestations) | 3
Infection with normal ANC - bladder (urinary) (Infections and infestations) | 4
Infection with normal ANC - pharynx (Infections and infestations) | 3
Infection with normal ANC - skin (cellulites) (Infections and infestations) | 3
Insomnia (General disorders) | 6
Irregular menses (Reproductive system and breast disorders) | 4
Left ventricular systolic function (Cardiac disorders) | 3
Leukocytes (Blood and lymphatic system disorders) | 14
Lymphopenia (Investigations) | 18
Mood Alteration (Psychiatric disorders) | 5
Mood alteration - anxiety (Psychiatric disorders) | 3
Mucositis (clinical exam) - oral cavity (Gastrointestinal disorders) | 13
Mucositis - oral cavity (Gastrointestinal disorders) | 32
Muscle weakness - whole body/generalized (General disorders) | 4
Nail changes (Skin and subcutaneous tissue disorders) | 7
Nausea (Gastrointestinal disorders) | 13
Neuropathy - motor (Nervous system disorders) | 3
Neuropathy - sensory (Nervous system disorders) | 7
Neutrophils (Blood and lymphatic system disorders) | 12
Pain - abdominal NOS (General disorders) | 6
Pain - back (General disorders) | 4
Pain - bone (General disorders) | 11
Pain - chest/thorax (General disorders) | 4
Pain - extremity-limb (General disorders) | 9
Pain - head/headache (General disorders) | 11
Pain - joint (General disorders) | 8
Pain - muscle (General disorders) | 11
Pain - oral cavity (General disorders) | 4
Pain - pain NOS (General disorders) | 4
Pain - throat/pharynx/larynx (General disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 10
Supraventricular arrhythmia - sinus tachycardia (Cardiac disorders) | 3
Sweating (General disorders) | 3
Taste alteration (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 10
Weight loss (General disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days